CLINICAL TRIAL: NCT06486519
Title: Collection of Vaginal Microbiota from Healthy Women Subject to Vaginal and Urinary Infections (VAGINOTYPE)
Brief Title: Collection of Vaginal Microbiota Samples (VAGINOTYPE)
Acronym: VAGINOTYPE
Status: Completed | Type: Observational
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Other Study IDs: L-031; 2022-A01997-36 (Other: ID-RCB)
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vaginal Microbiota
Keywords: VAGINOTYPE; Urinary tract infections; Vaginal infections; Women's health
MeSH Terms: conditions — Urinary Tract Infections; Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to collect vaginal microbiota samples from healthy women who are subject to vaginal and urinary infections.

DETAILED DESCRIPTION:
The goal of this study is to collect vaginal swab samples in order to gain knowledge on vaginal microbial communities of healthy women who have had experiences with vaginal and urinary infections.

Eligible participants will be enrolled in the study for a total duration of 1 day, where they will provide consent, answer a questionnaire and collect the vaginal samples.

ELIGIBILITY:
Inclusion Criteria:

I1. Age between 18 and 60 years (limits included),

I2. BMI between 18 and 30 kg/m² (limits included),

I3. Good general and mental health within the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,

I4. Able and willing to participate to the study by complying with the protocol procedures as evidenced by the dated and signed informed consent form,

I5. Affiliated with a social security scheme,

I6. Women who have had a vaginal or urinary infection in the last two years.

Exclusion Criteria:

E1. Suffering from gastrointestinal acute or chronic disease or complication (e.g. celiac disease, gastroesophageal reflux disease, gastric or duodenal ulcer, Crohn's disease, hemorrhoids, irritable bowel syndrome) or frequent gastrointestinal disorders (e.g. diarrhea, nausea, vomiting, abdominal pain, constipation, hemorrhoids...)

E2. Any infectious gastrointestinal complaint within 4 weeks before V1

E3. Suffering from a metabolic disorder such as diabetes, thyroidal trouble, arterial hypertension or other metabolic disorder or any disease requiring a chronic treatment

E4. Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, cardiac, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or disease found to be inconsistent with the conduct of the study by the investigator

E5. Suffering from a pathology of the oral sphere (untreated caries, gingivitis, periodontitis, abscess, etc.) or having a positive result in an oral swab test for STIs (chlamydia, gonococcus, syphilis, herpes, etc.)

E6. Women affected by a Sexually Transmitted Infection (STI) or Disease (STD) such as HPV (Human PapillomaVirus), Chlamydia infection, syphilis, gonorrhea, genital herpes

E7. Having undergone a surgical procedure likely to disrupt the gut microbiome within the 6 months prior to the V1 visit, especially bariatric surgery

E8. Coloscopy within 3 months prior to the visit

E9. Women who gave birth within one year of the visit, women who are pregnant or intend to become pregnant during the study, women who are breastfeeding

E10.Previous or current antibiotic, antiviral, antifungal, proton pump inhibitor, or any treatment which may disrupt the microbiota in the 4 weeks prior to the V1 visit

E11.In the process of quitting smoking or having started smoking less than 6 months ago

E12.Taking part in another clinical trial or being in the exclusion period of a previous clinical trial

E13. Having received, during the last 12 months, indemnities for clinical trial higher or equal to 6000 Euros

E14.Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision

E15.Presenting a psychological or linguistic incapability to sign the informed consent

E16.Impossible to contact in case of emergency

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy females from 18 to 60 years of age inclusively that are willing to participate in the study and to provide a vaginal swab sample. Females that are subject to vaginal or urinary infections.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Composition of the vaginal microbiome | 1 day
  Vaginal microbiota composition (α-diversity, β-diversity, and relative abundance at the genus and species level) at a single point in time via shotgun sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Metreau, MD, Principal Investigator — Biofortis, Unité d'Investigation Clinique de Saint-Herblain
Locations (2):
- France (2):
  - Biofortis, Unité d'Investigation Clinique, Paris
  - Biofortis, Unité d'Investigation Clinique, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No